CLINICAL TRIAL: NCT02884635
Title: Phase IIa Study of ASP1707 A Randomized, Placebo-Controlled, Double-Blind, Parallel Group Phase 2a Study of ASP1707 in Postmenopausal Female Patients With Rheumatoid Arthritis (RA) Taking Methotrexate (MTX)
Brief Title: A Study to Evaluate the Efficacy and Safety of ASP1707 in Postmenopausal Female Patients With Rheumatoid Arthritis Taking Methotrexate
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1707-CL-3001
Record Dates: First submitted 2016-08-26; First posted 2016-08-31 (Estimated); Last update posted 2024-10-23 (Actual); Status verified 2024-10

CONDITIONS: Rheumatoid Arthritis
Keywords: Methotrexate; ASP1707; Rheumatoid arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — opigolix; Methotrexate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ASP1707 (Experimental): ASP1707 will be orally administered for 12 weeks.
  Interventions: Drug: ASP1707; Drug: Methotrexate
- Placebo (Placebo Comparator): Placebo will be orally administered for 12 weeks.
  Interventions: Drug: Placebo; Drug: Methotrexate

INTERVENTIONS:
Drug: ASP1707 — Oral
  Arms: ASP1707
Drug: Placebo — Oral
  Arms: Placebo
Drug: Methotrexate — Methotrexate will be orally administered at stable dose from at least 28 days prior to screening through the screening and treatment periods until the end of the follow-up period.

SUMMARY:
The objective of this study is to evaluate the efficacy, pharmacokinetics, pharmacodynamics and safety of ASP1707 in combination with MTX in postmenopausal female patients with RA.

ELIGIBILITY:
Inclusion Criteria:

* Subject has RA that was diagnosed according to the 1987 ACR criteria or the 2010 ACR/EULAR criteria.
* Subject meets the ACR 1991 Revised Criteria for the Classification of Global Functional Status in RA Class I, II or, III.
* subject has active RA as evidenced by both of the followings:

  * ≥ 6 tender/painful joints (using 68-joint assessment)
  * ≥ 6 swollen joints (using 66-joint assessment)
* CRP (C-reactive protein) of > 0.3 mg/dL or ESR (Erythrocyte sedimentation rate) of > 28 mm/hr at screening.
* Subject who continuously received MTX and who is able to continue stable dose of MTX.
* Subject who did not receive the following drugs, or received the drugs with stable dosage:

Non-steroidal anti-inflammatory drugs, oral morphine or equivalent opioid analgesics, acetaminophen, or oral corticosteroids.

Exclusion Criteria:

* Inadequate responders to a biologic DMARD (Disease-modifying antirheumatic drug).
* Subject has taken other investigational research products are prohibited within 12 weeks (84 days) or within 5 half-lives, whichever is longer, prior to screening.
* Subject has undergone surgery which has residual effects on the assessed joints, or is scheduled to undergo surgery that may affect the study evaluation of the assessed joints.
* Subject has another type of inflammatory arthritis other than RA.
* Subject who meets any of the following criteria of laboratory values at screening:

  * White blood cell count <4000/μL
  * Platelet count <100000/μL
  * ALT (Alanine Aminotransferase) ≥ 2 x ULN (Upper Limit of Normal)
  * AST (Aspartate Aminotransferase) ≥ 2 x ULN
  * Total bilirubin ≥ 1.5 x ULN
  * Positive Hepatitis B surface antigen, Hepatitis B virus-DNA quantitation, or Hepatitis C virus antibody
* Subject has a positive QuantiFERON-TB Gold test or T-spot.
* Subject has a history of or concurrent malignant tumor.
* Subject has any ongoing severe, progressive, or uncontrolled renal, hepatic, hematological, gastrointestinal, metabolic, endocrine, pulmonary, cardiac, neurological, infectious, or autoimmune disease except for RA, or diseases which preclude the subject's participation in the study.
* Subject has a history of clinically significant allergy.
* Subject has clinically significant abnormalities on the 12-lead Electrocardiogram.
* Subject has a history of positive Human Immunodeficiency Virus infection.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2016-09-16 (Actual); Primary Completion 2017-10-18 (Actual); Study Completion 2017-10-25 (Actual)

PRIMARY OUTCOMES:
ACR20 response rate | Week 12
  ACR20: American College of Rheumatology 20

SECONDARY OUTCOMES:
ACR20 response rate | Up to Week 8
ACR50 response rate | Up to Week 12
ACR70 response rate | Up to Week 12
Change from baseline in DAS28-CRP score | Baseline and Up to Week 12
  DAS28-CRP: Disease Activity Score28 - C-reactive protein
Change from baseline in DAS28-ESR score | Baseline and Up to Week 12
  DAS28-ESR: Disease Activity Score28 - Erythrocyte sedimentation rate
Change from baseline in Tender Joint Count (68 joints) | Baseline and Up to Week 12
Change from baseline in Swollen Joint Count (66 joints) | Baseline and Up to Week 12
Percentage of subjects achieving DAS28-CRP score and DAS28-ESR score for remission (<2.6) | Up to Week 12
Percentage of subjects achieving DAS28-CRP score and DAS28-ESR score for low disease activity (≤3.2) | Up to Week 12
Change from baseline in CRP | Baseline and Up to Week 12
Change from baseline in ESR | Baseline and Up to Week 12
Percentage of subjects achieving EULAR response criterion of "Good Response" | Up to Week 12
  EULAR: European league Against Rheumatism
Percentage of subjects achieving EULAR response criterion of "Good Response" or "Moderate Response" | Up to Week 12
Percentage of subjects achieving ACR/EULAR score for remission | Up to Week 12
Percentage of subjects achieving SDAI score ≦ 3.3 (SDAI remission) | Up to Week 12
  SDAI: Simplified Disease Activity Index
Change from baseline in the SDAI score | Baseline and Up to Week 12
Change from baseline for the HAQ-DI | Baseline and Up to Week 12
  HAQ-DI: Health Assessment Questionnaire - Disability Index
Safety assessed by incidence of adverse events | Up to Week 13
Safety assessed by body temperature | Up to Week 13
Safety assessed by pulse rate | Up to Week 13
Safety assessed by blood pressure in sitting position | Up to Week 13
Safety assessed by laboratory tests: Hematology | Up to Week 13
Safety assessed by laboratory tests: Biochemistry | Up to Week 13
Safety assessed by laboratory tests: Urinalysis | Up to Week 13
Safety assessed by standard 12-lead electrocardiogram | Up to Week 13
Safety assessed by weight | Up to Week 13
Plasma concentration of ASP1707 | Up to Week 12
Plasma concentration of metabolite of ASP1707 | Up to Week 12
Pharmacodynamics assessed by endocrinology tests | Up to Week 13
Pharmacodynamics assessed by plasma concentration of TNF-α | Up to Week 13
  TNF: Tumor Necrosis Factor
Pharmacodynamics assessed by plasma concentration of MMP3 | Up to Week 13
  MMP3: Matrix metalloproteinase 3
Pharmacodynamics assessed by plasma concentration of IL-6 | Up to Week 13
  IL-6: Interleukin-6

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Astellas Pharma Inc
Locations (27):
- Japan (27):
  - Site JP00004, Numakunai, Iwate
  - Site JP00005, Numakunai, Iwate
  - Site JP00022, Aichi
  - Site JP00023, Aichi
  - Site JP00017, Chiba
  - Site JP00026, Ehime
  - Site JP00025, Fukui
  - Site JP00012, Fukuoka
  - Site JP00018, Fukuoka
  - Site JP00019, Fukuoka
  - Site JP00006, Gunma
  - Site JP00024, Gunma
  - Site JP00010, Hiroshima
  - Site JP00011, Hiroshima
  - Site JP00001, Hokkaido
  - Site JP00002, Hokkaido
  - Site JP00003, Hokkaido
  - Site JP00016, Kagoshima
  - Site JP00007, Kanagawa
  - Site JP00021, Kanagawa
  - Site JP00014, Kumamoto
  - Site JP00015, Kumamoto
  - Site JP00013, Nagasaki
  - Site JP00020, Ōita
  - Site JP00008, Shizuoka
  - Site JP00009, Shizuoka
  - Site JP00027, Tokyo

IPD SHARING:
Plan to Share IPD: Yes
Access to anonymized individual participant level data collected during the study, in addition to study-related supporting documentation, is planned for studies conducted with approved product indications and formulations, as well as products terminated during development. Studies conducted with product indications or formulations that remain active in development are assessed after study completion to determine if Individual Participant Data can be shared. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Access to participant level data is offered to researchers after publication of the primary manuscript (if applicable) and is available as long as Astellas has legal authority to provide the data.
Access Criteria: Researchers must submit a proposal to conduct a scientifically relevant analysis of the study data. The research proposal is reviewed by an Independent Research Panel. If the proposal is approved, access to the study data is provided in a secure data sharing environment after receipt of a signed Data Sharing
URL: https://www.clinicaltrials.astellas.com/transparency/

REFERENCES:
- See also: Link to results on the Astellas Clinical Study Results website — https://www.astellasclinicalstudyresults.com/hcp/findresult.aspx?RID=;;;1707-CL-3001;;;